CLINICAL TRIAL: NCT01811576
Title: A 64-Week (12-week Core Phase and 52-week Safety Extension), Phase II, Multicenter, Randomized, Open Label Study to Evaluate the Safety, Tolerability and Efficacy of Weekly TV-1106 in Adults With Growth Hormone Deficiency
Brief Title: Safety, Tolerability and Efficacy of Weekly TV-1106 in Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV1106-GHD-201; 2012-004975-37 (EudraCT Number)
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth hormone deficiency; Insulin-like growth factor I (IGF-I); TV-1106
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — albusomatropin; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- recombinant human growth hormone (Active Comparator): Daily subcutaneous dose
  Interventions: Drug: Recombinant human growth hormone
- TV-1106 (Experimental): Titration dose levels of TV-1106
  Interventions: Drug: TV-1106

INTERVENTIONS:
Drug: TV-1106
  Arms: TV-1106
Drug: Recombinant human growth hormone — Subcutaneous once daily
  Arms: recombinant human growth hormone

SUMMARY:
The primary objective of this study is to evaluate the clinical effect of TV-1106.

ELIGIBILITY:
Inclusion Criteria:

* Patient agrees to provide written informed consent and to comply with the study protocol after reading the informed consent and discussing the study with the investigator.
* Males and females between 23 and 65 years of age must have a confirmed diagnosis of adult GHD, either adult onset (AO) GHD due to hypothalamic-pituitary disease or childhood onset (CO) GHD that is either idiopathic or due to hypothalamic-pituitary disease or due to genetic causes.
* Diagnosis of GH deficiency must be confirmed by documented (medical records) diagnostic testing.
* Patients should have been treated with a stable dose of daily rhGH for at least 3 months prior to screening.
* Other criteria apply.

Exclusion Criteria:

* Patients with history or clinical evidence of active or chronic diseases that could confound results of the study or put the subject at undue risk as determined by the investigator.
* Patients with known active malignancy
* Patients with history of malignancy other than intracranial tumor causing GHD (excluding surgically cured basal cell or squamous cell cancer of the skin with documented 6 month remission)
* Patients with evidence of pituitary adenoma or other intracranial tumor within 12 months of enrollment, which is on day 0 (baseline, Visit 3)
* Patients without magnetic resonance imaging (MRI) or computerized tomography (CT) data to document tumor stability within the 12 months prior to enrollment, which is on day 0 (baseline, Visit 3)
* Presence of Prader-Willi syndrome, Turner's syndrome, untreated adrenal insufficiency, active acromegaly in the past 5 years, or active Cushing's syndrome in the past 1 year.
* Other criteria apply.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03-31 (Actual); Primary Completion 2013-08-05 (Actual); Study Completion 2013-08-05 (Actual)

PRIMARY OUTCOMES:
Insulin-like growth factor I (IGF-I) concentration change from baseline | Baseline to Week 12

SECONDARY OUTCOMES:
Percentage of patients treated with TV1106 who return to pre-treatment IGF-1 SDS | Baseline to Week 12
Safety Parameters | 78 weeks
  The safety of TV-1106 will be assessed throughout the study by evaluating adverse events,concomitant medication usage, physical examinations including urinalysis and body weight, vital sign measurements, clinical laboratory test results and hormone levels, electrocardiograms (ECGs), and immunogenicity.

CONTACTS AND LOCATIONS:
Locations (23):
- Teva Investigational Site 10564, Portland, Oregon, United States
- Czechia (2):
  - Teva Investigational Site 54052, Hradec Králové
  - Teva Investigational Site 54051, Olomouc
- Germany (3):
  - Teva Investigational Site 32239, Dresden
  - Teva Investigational Site 32238, Munich
  - Teva Investigational Site 32237, Munich
- Greece (2):
  - Teva Investigational Site 63044, Athens
  - Teva Investigational Site 63045, Athens
- Hungary (7):
  - Teva Investigational Site 51056, Budapest
  - Teva Investigational Site 51055, Budapest
  - Teva Investigational Site 51060, Debrecen
  - Teva Investigational Site 51061, Győr
  - Teva Investigational Site 51059, Pécs
  - Teva Investigational Site 51057, Szeged
  - Teva Investigational Site 51058, Szolnok
- Israel (3):
  - Teva Investigational Site 80033, Jerusalem
  - Teva Investigational Site 80032, Petah Tikva
  - Teva Investigational Site 80034, Tel Aviv
- Teva Investigational Site 61029, Belgrade, Serbia
- Slovakia (3):
  - Teva Investigational Site 62017, Bratislava
  - Teva Investigational Site 62022, Bratislava
  - Teva Investigational Site 62016, Ľubochňa
- Teva Investigational Site 64016, Ljubljana, Slovenia